CLINICAL TRIAL: NCT01937078
Title: An 'N-of-1' Study of the Histamine H@ Antagonist, Famotidine in Levodopa-induced Dyskinesia in Parkinson's Disease
Brief Title: Famotidine for Levodopa-induced Dyskinesia in PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Susan Fox, PI, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDC FAM 2010
Record Dates: First submitted 2012-07-26; First posted 2013-09-09 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Dyskinesia
MeSH Terms: conditions — Dyskinesias | interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- active (Active Comparator): Famotidine will be administered at total daily doses of 80, 120mg, or 160mg per day. Each patient will be randomized to receive each active dose of famotidine (80, 120, or 160mg/d and placebo). Each patient will receive 4 randomized treatment phases - three famotidine (one at each of the dose levels) and one placebo.
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Famotidine — Each patient will receive 4 randomized treatment phases - three famotidine (one at each of the dose levels) and one placebo. Each treatment phase will last for 14 days. Doses of drug will be titrated upwards, starting at 40mg once daily on day one, 40mg twice daily on day two, and 80mg twice daily (or placebo + drug equivalent) from day three and then continue on this dose for the next 12 days. Regardless of treatment phase, subjects will take 2 tablets twice daily, with varying ratios of active famotidine to placebo. Thus famotidine 80mg/d will consist of 1 tablet of 40 mg famotidine plus 1 tablet of placebo twice a day; 120 mg /d famotidine will be 2 tablets at 40 mg morning and 1 tablet famotidine 40 mg plus 1 tablet placebo evening; famotidine 160 mg/d will be famotidine 40 mg tablets, 2 tablets twice a day. The placebo phase will consist of 2 placebo tablets twice a day.

SUMMARY:
Levodopa-induced dyskinesia is a common problem in Parkinson's disease (PD). In particular, targeting non-dopaminergic systems may be an option for reducing dyskinesia without worsening motor symptoms. One such target may be histamine. The central histaminergic system is involved in diverse biological functions including thermoregulation, eating, and sleep; a role in motor activity is suggested by strong histaminergic innervation of the basal ganglia. Histamine H2 receptors are highly expressed in the striatum, particularly on the GABAergic striatal-pallidal and striatal-nigral pathways Histamine H2 stimulation modulates acetylcholine release. Previous studies have demonstrated that blocking acetylcholine with anticholinergic agents can induce chorea. The investigators propose that histamine H2 receptor stimulation decreases acetylcholine in the striatum and increases activity of the direct striatal output pathway, a key component of the neural mechanisms underlying dyskinesia.

The investigators hypothesise that H2 antagonists would reduce activity of the direct striatopallidal pathway and so potentially reduce levodopa-induced chorea

Famotidine has also been assessed in schizophrenia in a small cases series to treat schizophrenia, with tolerability. Clinical experience thus suggests the suitability of using this agent as a histamine H2 antagonist in clinical studies for PD.

DETAILED DESCRIPTION:
The proposed study will be composed of multiple N -of 1 studies performed in a randomized, double-blind, placebo-controlled multiple (4) crossover fashion. Twelve PD patients (thus 12 N-of-1 trials) with levodopa-induced dyskinesia will complete 4 treatment phases; one phase at each of the 3 doses of famotidine and one of placebo. The treatment doses will be: famotidine 40mg/day, 80mg/day, and 120mg/day. The phases will occur in a random order, but each subject will receive each of the treatment doses during the course of the study. After each phase of treatment (14 days), there will be a washout period (7 days, over 10 half-lives of famotidine) followed by a crossover. The primary outcome will be the change in Unified Dyskinesia Rating Scale (UDysRS) between placebo and famotidine at the end of each treatment phase and secondary outcomes will be Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) parts III and IV, Clinical Global Impression (CGI), Lang-Fahn activities of daily living dyskinesia scale (LFADLDS) and assessment of adverse effects.

ELIGIBILITY:
Inclusion Criteria:Eligible patients, male and female, will be less than 80 years of age and be on stable levodopa. Subjects must have stable, bothersome dyskinesia and have an MDS-UPDRS score 2 or greater, on item 4.2. All anti-parkinsonian medications must be unchanged for at least one month prior to study enrollment. Subjects may be taking amantadine at a stable dose for at least one month prior to study onset -

Exclusion Criteria:are prior surgery for PD, Hoehn and Yahr score of 5 when off-medication, history of moderate to severe renal impairment (creatinine clearance <25 millilitres per minute, dementia (defined by Montreal Cognitive Scale < 2518 , allergic reaction to lactose, famotidine or other histamine H2 antagonists

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Dyskinesia severity using Unified Dyskinesia Rating Scale | on days 1;14;21;35;42;56;63;77

SECONDARY OUTCOMES:
Subject-rated dyskinesia severity using Unified Dyskinesia Rating Scale and Lang-Fahn Activities of Daily Living Scale | on days 1;14;21;35;42;56;63;77
Parkinsonian disability using UPDRS (blinded investigator-rated | on days 1;14;21;35;42;56;63;77
Adverse events | on days 1;14;21;35;42;56;63;77
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Susan Fox, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada